CLINICAL TRIAL: NCT00223145
Title: Randomized, Multicentre, Phase III Study in Patients With Intermediate-risk T1 T2 Prostate Adenocarcinomas, to Verify the Role of Six Months of Total Androgen Blockade for Two Dosage Levels of Prostate Radiation Therapy (70 Gy and 76 Gy) Versus Prostate Radiation Therapy Alone at 76 Gy
Brief Title: Study on the Role of Hormonal Treatment for Two Dosage Levels of Prostate Radiation Therapy Versus Prostate Radiation Therapy Alone
Acronym: PCS III
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abdenour Nabid (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Abdenour Nabid, Principal Investigator, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-990-0049,1; DC-990-0049
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate adenocarcinoma; Gleason score <= 6 and PSA 10-20; Gleason score = 7 and PSA <=20
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Androgen blockade for 6 months + Radiotherapy 70 Gy
  Interventions: Radiation: Radiotherapy 70 Gy; Drug: Androgen blockade
- Arm 2 (Experimental): Androgen blockade for 6 months + Radiotherapy 76 Gy
  Interventions: Radiation: Radiotherapy 76 Gy; Drug: Androgen blockade
- Arm 3 (Active Comparator): Radiotherapy alone with 76 Gy
  Interventions: Radiation: Radiotherapy 76 Gy

INTERVENTIONS:
Radiation: Radiotherapy 70 Gy — Radiotherapy to the prostate
  Arms: Arm 1
Radiation: Radiotherapy 76 Gy — Radiotherapy to the prostate
  Arms: Arm 2; Arm 3
Drug: Androgen blockade — Duration : 6 months
  Other Names: Bicalutamide 50 mg; Goserelin 10.8 mg
  Arms: Arm 1; Arm 2

SUMMARY:
The hypothesis of the proposed study would be that, due to the six months of total androgen blockade, which would include neoadjuvant hormonal therapy for four months and concomitant hormonal therapy for two months with irradiation, the investigators could reduce local failure rates for these two dosage levels, namely 70 Gy and 76 Gy. Since increasing the dose to the prostate also seems to reduce local relapse rates, the results of the two hormonal therapy groups would be compared with the results of prostate irradiation at doses of 76 Gy. This study would verify the possibility of compensating a six Gy dosage increase of radiation therapy with six months of hormonal therapy between the 70 Gy and 76 Gy groups who received hormonal therapy, and also match these results with a dose escalation to the prostate of 76 Gy. In the future, this could result in more therapeutic choices, such as reducing the doses of radiation therapy and, consequently, its related complications, if hormonal therapy proves to be beneficial; or rather, to continue in the direction of dose escalation for this intermediate-risk patient group, everything being correlated to the side effects of hormonal therapy and irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage T1 or T2 untreated adenocarcinoma of the prostate, with a Gleason score that is less than or equal to 6, as well as a prostate-specific antigen (PSA) between 10-20 (intermediate risk) or patients with stage T1 or T2 untreated adenocarcinoma of the prostate, with a Gleason score that is equal to 7, as well as a PSA equal to or less than 20 (intermediate risk).
* Performance status score of 0-1
* Patients must sign a consent form before starting the study.
* No evidence of regional disease
* Patients with a previous history of cancer are eligible on the condition that they have been disease-free for more than five years.
* Non-invasive epidermoid cancers of the skin are eligible.
* The patient must be available for treatments and follow-up visits.
* No evidence of metastatic disease, confirmed by a negative bone scan.

Exclusion Criteria:

* Severe medical or psychiatric problems that may compromise study compliance
* Chronic hepatic disease; abnormal hepatic function, i.e. aspartate aminotransferase and alanine aminotransferase > 1.5 times the upper normal limit.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2000-12; Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Interval before biochemical failure | 10 years

SECONDARY OUTCOMES:
Toxicity of irradiation | 10 years
Survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Abdenour Nabid, MD, Principal Investigator — CRC - CHUS
Locations (1):
- Centre de Recherche Clinique du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Nabid A, Carrier N, Vigneault E, Van Nguyen T, Vavassis P, Brassard MA, Bahoric B, Archambault R, Vincent F, Bettahar R, Wilke D, Souhami L. Androgen deprivation therapy and radiotherapy in intermediate-risk prostate cancer: A randomised phase III trial. Eur J Cancer. 2021 Jan;143:64-74. doi: 10.1016/j.ejca.2020.10.023. Epub 2020 Dec 3. PMID 33279855